CLINICAL TRIAL: NCT03704350
Title: Influence of Obesity on Endogenous Oxalate Synthesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Dean Assimos, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300002318-P20; P20DK119788 (NIH); UAB (Other: UAB)
Record Dates: First submitted 2018-10-03; First posted 2018-10-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 20-24.9 BMI (Active Comparator): Participants with a BMI that falls between 20 and 24.9 who will receive the controlled diet
  Interventions: Dietary Supplement: controlled diet
- 25-29.9 BMI (Active Comparator): Participants with a BMI that falls between 25 and 29.9 who will receive the controlled diet
  Interventions: Dietary Supplement: controlled diet
- 30-34.9 BMI (Active Comparator): Participants with a BMI that falls between 30 and 34.9 who will receive the controlled diet
  Interventions: Dietary Supplement: controlled diet
- 35-39.9 BMI (Active Comparator): Participants with a BMI that falls between 35 and 39.9 who will receive the controlled diet
  Interventions: Dietary Supplement: controlled diet
- 40-44.9 BMI (Active Comparator): Participants with a BMI that falls between 40 and 44.9 who will receive the controlled diet
  Interventions: Dietary Supplement: controlled diet
- 45-50 BMI (Active Comparator): Participants with a BMI that falls between 45 and 50 who will receive the controlled diet.
  Interventions: Dietary Supplement: controlled diet

INTERVENTIONS:
Dietary Supplement: controlled diet — Participants will consume a diet that is controlled in its daily contents of oxalate, calcium, vitamin C and sodium, and in its content of carbohydrate, fat, and protein. Participants will be asked not to take any dietary supplements (vitamins, calcium or other minerals, herbal supplements, nutritional aids), to exercise strenuously, or to consume food or drink that is not provided to them as part of the controlled diet.

SUMMARY:
There is increasing evidence that obesity is associated with increased urinary oxalate excretion, an important risk factor for calcium oxalate stone formation. By the administration of a controlled low oxalate diet the investigators will estimate endogenous oxalate synthesis in both non-obese and obese non-kidney-stone forming adults. This study seeks to thusly increase the understanding of the relationships between obesity and endogenous oxalate synthesis to serve as a platform to develop novel therapies for stone prevention.

DETAILED DESCRIPTION:
Calcium oxalate stone disease results in billions of dollars in healthcare costs per year, creates large economic losses due to decreased work productivity, and produces significant pain and suffering in affected individuals impacting quality of life. Almost 9% of the population in the United States may now experience a stone event at least once in their lifetime and that figure is increasing. Although stone removing treatments have advanced in the last few decades with a variety of minimally invasive procedures such as shock wave lithotripsy, ureteroscopy and percutaneous nephrolithotomy, our knowledge of how stones form and how to prevent them has not kept pace. Approximately 70-80% of the stones formed contain oxalate. Oxalate is an end product of metabolism and an ubiquitous element of human diets. Small increases in urinary oxalate can increase calcium oxalate crystal formation and thus stone disease. Urinary oxalate levels are affected by both dietary and endogenous components, complicating the discrimination between the two sources. Multiple epidemiological and clinical studies have demonstrated a link between body mass index (BMI) and kidney stone disease and also an increased urinary oxalate excretion.

The interpretation of studies suggesting a link between obesity and the amount of urinary oxalate excreted is confounded by the failure in most studies to use diets controlled in calcium and oxalate. Adult humans without a history of kidney stones will be placed on controlled low oxalate diets to estimate the contribution of endogenous oxalate synthesis to the urinary oxalate pool. In addition, oral doses of 13C2-glycolate and 13C6- vitamin C will be used to determine their conversions to 13C2-oxalate and provide an index of endogenous oxalate production. Body morphometric indices, markers of oxidative stress, and insulin resistance will be assessed in these subjects.They will also be evaluated with DXA and MRI to define body fat content and distribution.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-60 years
* Body Mass Index (BMI) <50

Exclusion Criteria:

* history of kidney stones
* history of diabetes, hepatic disease, renal disease including Chronic Kidney Disease (CKD), bowel disease or other endocrine disorders
* pregnant or lactating women, or those with the intention to become pregnant in the near future
* abnormal liver enzymes
* hemoglobin A1C > 6.5

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-24 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Urinary oxalate excretion | Baseline through Day 12
  Urinary oxalate excretion from 24 hour urine collections will be reported as mg/day.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Assimos, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No